CLINICAL TRIAL: NCT02933879
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Multi- Site Phase 2b Clinical Study to Assess the Efficacy, Safety and Tolerability Patients With Mild to Moderate Onychomycosis
Brief Title: Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Multi-Site Phase 2b Clinical Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVXT 1404
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Results first posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVXT topical (Experimental): daily dosing for one 8-week treatment period (Treatment Group A) and two 8-week treatment periods separated by a 32-week rest period (Treatment Group B),
  Interventions: Drug: NVXT topical
- Placebo (Vehicle) Topical (Placebo Comparator): two 8-week treatment periods separated by a 32-week rest period (Treatment Group C),
  Interventions: Drug: Placebo (Vehicle) Topical

INTERVENTIONS:
Drug: NVXT topical — topical treatment
  Other Names: Active
  Arms: NVXT topical
Drug: Placebo (Vehicle) Topical — Placebo (Vehicle) Topical
  Other Names: placebo
  Arms: Placebo (Vehicle) Topical

SUMMARY:
A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group, Multi- Site Phase 2b Clinical Study to Assess the Efficacy, Safety and Tolerability of 8-Week Regimens of NVXT topical product in Patients with Mild to Moderate Onychomycosis

DETAILED DESCRIPTION:
Evaluate safety and tolerability of the two regimens of NVXT (Treatment Groups A and B) in patients with mild to moderate distal subungual onychomycosis of the target toenail.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of onychomycosis of the target toenail (defined as one of the infected great toenails).

Exclusion Criteria:

* Females who are pregnant, lactating or likely to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Novum Pharmaceutical Research Services (Novum), Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NVXT Topical Treatment Group A: daily dosing for one 8-week treatment period
  NVXT topical: topical treatment
- NVXT Topical Treatment Group B: daily dosing for two 8-week treatment periods separated by a 32-week rest period
  NVXT topical: topical treatment
- Placebo (Vehicle) Topical Treatment Group C: two 8-week treatment periods separated by a 32-week rest period
  Placebo (Vehicle) Topical: Placebo (Vehicle) Topical
Period: Overall Study
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C
Started | 64 | 62 | 58
Completed | 48 | 48 | 41
Not Completed | 16 | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C | Total
Number analyzed (Participants) | 64 | 62 | 58 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (15.0) | 53.1 (14.7) | 50.8 (12.6) | 51.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 21 | 59
  Male | 43 | 45 | 37 | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 38 | 39 | 118
  Not Hispanic or Latino | 23 | 24 | 19 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 7 | 8 | 27
  White | 52 | 55 | 50 | 157
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Treatment Group With a Complete Therapeutic Cure
Description: Complete therapeutic cure is defined as both complete clinical and mycological cure of the target toenail
Time Frame: Day 365
Population: 1 Subject from Group B and 1 Subject from Group C were excluded from Efficacy Analysis because they did not have positive mycological culture screenings. Also, 12 subjects from Group A, 13 from Group B, and 14 from Group C were excluded because they had no efficacy data for the relevant analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 52 | 48 | 43
Participants | 1 | 0 | 1
Statistical Analysis 1: Comparison: NVXT Topical Treatment Group B vs Placebo (Vehicle) Topical Treatment Group C; Test type: Superiority; p = 0.4615, Z-test, 2 sided

2. Primary Outcome: Number of Patients in Each Treatment Group With a Complete Therapeutic Cure
Description: Complete therapeutic cure is defined as both complete clinical and mycological cure of the target toenail
Time Frame: Day 141
Population: Groups A and B were combined to compare against Group C to determine statistically significant difference when combining both groups that received test treatment in the first 56 Days vs only placebo. 19 subjects from Group A+B and 9 from Group C were excluded because they had no efficacy data or they lacked positive mycological cultures.
Measure: Count of Participants; unit: Participants
Groups:
- NVXT Topical Treatment Group A+B: daily dosing for one 8-week treatment period (Treatment Group A) and two 8-week treatment periods separated by a 32-week rest period (Treatment Group B),
  NVXT topical: topical treatment
- Placebo (Vehicle) Topical Treatment Group C: two 8-week treatment periods separated by a 32-week rest period (Treatment Group C),
  Placebo (Vehicle) Topical: Placebo (Vehicle) Topical
Arm/Group | NVXT Topical Treatment Group A+B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 107 | 49
Participants | 0 | 1

3. Secondary Outcome: Number of Patients in Each Treatment Group With a Complete or Almost Complete Therapeutic Cure
Description: Almost complete therapeutic cure is defined as both mycological and satisfactory clinical cure of the target toenail
Time Frame: Day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 52 | 48 | 43
Participants | 2 | 2 | 4
Statistical Analysis 1: Comparison: NVXT Topical Treatment Group B vs Placebo (Vehicle) Topical Treatment Group C; Test type: Superiority; p = 0.0404, Z-test, 2 sided
Statistical Analysis 2: Comparison: NVXT Topical Treatment Group A vs Placebo (Vehicle) Topical Treatment Group C; Test type: Superiority; p = 0.2106, Z-test, 2 sided

4. Secondary Outcome: Number of Patients in Each Treatment Group With a Complete or Almost Complete Therapeutic Cure
Description: Almost complete therapeutic cure is defined as both mycological and satisfactory clinical cure of the target toenail
Time Frame: Day 141
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A+B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 107 | 49
Participants | 1 | 1

5. Secondary Outcome: Number of Patients in Each Treatment Group With a Mycological Cure
Description: Mycological cure is defined as a negative KOH test and a negative fungal culture.
Time Frame: day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 52 | 48 | 43
Participants | 7 | 13 | 12
Statistical Analysis 1: Comparison: NVXT Topical Treatment Group B vs Placebo (Vehicle) Topical Treatment Group C; Test type: Superiority; p = 1.0000, Z-test, 2 sided

6. Secondary Outcome: Number of Patients in Each Treatment Group With a Mycological Cure
Description: Mycological cure is defined as a negative KOH test and a negative fungal culture.
Time Frame: Day 141
Population: Groups A and B were combined to compare against Group C to determine statistically significant difference when combining both groups that received test treatment in the first 56 Days vs only placebo. 20 subjects from Group A+B and 10 from Group C were excluded because they had no efficacy data or they lacked positive mycological cultures.
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A+B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 106 | 48
Participants | 30 | 10

7. Secondary Outcome: Number of Patients in Each Treatment Group With a Complete Clinical Cure
Description: Complete clinical cure is defined as 0% nail involvement.
Time Frame: day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 52 | 48 | 43
Participants | 1 | 1 | 1
Statistical Analysis 1: Comparison: NVXT Topical Treatment Group B vs Placebo (Vehicle) Topical Treatment Group C; Test type: Superiority; p = 1.0000, Z-test, 2 sided

8. Secondary Outcome: Number of Patients in Each Treatment Group With a Complete Clinical Cure
Description: Complete clinical cure is defined as 0% nail involvement.
Time Frame: Day 281
Population: Groups A and B were combined to compare against Group C to determine statistically significant difference when combining both groups that received test treatment in the first 56 Days vs only placebo. 24 subjects from Group A+B and 15 from Group C were excluded because they had no efficacy data or they lacked positive mycological cultures.
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A+B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 102 | 43
Participants | 0 | 0

9. Secondary Outcome: Number of Patients in Each Treatment Group With a Complete Clinical Cure
Description: Complete clinical cure is defined as 0% nail involvement.
Time Frame: Day 141
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A+B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 107 | 49
Participants | 0 | 1

10. Secondary Outcome: Number of Patients in Each Treatment Group With a Satisfactory Clinical Cure
Description: Satisfactory clinical cure is defined as <5% of the target toenail involvement.
Time Frame: day 365
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 52 | 48 | 43
Participants | 7 | 2 | 5
Statistical Analysis 1: Comparison: NVXT Topical Treatment Group B vs Placebo (Vehicle) Topical Treatment Group C; Test type: Superiority; p = 0.2467, Z-test, 2 sided

11. Secondary Outcome: Number of Patients in Each Treatment Group With a Satisfactory Clinical Cure
Description: Satisfactory clinical cure is defined as <5% of the target toenail involvement.
Time Frame: Day 281
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A+B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 102 | 43
Participants | 2 | 1

12. Secondary Outcome: Number of Patients in Each Treatment Group With a Satisfactory Clinical Cure
Description: Satisfactory clinical cure is defined as <5% of the target toenail involvement.
Time Frame: Day 141
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NVXT Topical Treatment Group A+B | Placebo (Vehicle) Topical Treatment Group C
Number analyzed (Participants) | 107 | 49
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | NVXT Topical Treatment Group A | NVXT Topical Treatment Group B | Placebo (Vehicle) Topical Treatment Group C
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/62 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/62 | 1/58
Other Adverse Events (participants affected / at risk) | 19/64 | 14/62 | 13/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVXT Topical Treatment Group A (N=64) | NVXT Topical Treatment Group B (N=62) | Placebo (Vehicle) Topical Treatment Group C (N=58)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVXT Topical Treatment Group A (N=64) | NVXT Topical Treatment Group B (N=62) | Placebo (Vehicle) Topical Treatment Group C (N=58)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting projectile (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 0 (0) | 2 (2)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 4 (5) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Scrotal varicose veins (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT02933879/SAP_000.pdf
  • Study Protocol (2016-07-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT02933879/Prot_001.pdf